CLINICAL TRIAL: NCT03492619
Title: Intervention for Women in Costa Rica Who Are Discouraged and Have Food Insecurity and Excess Body Weight
Brief Title: Intervention for Women in Costa Rica
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Universidad de Costa Rica (Other); Municipality of Alajuela (Unknown); Agenda de Mujeres (Unknown)
Responsible Party: Principal Investigator, Edward Frongillo, Jr., Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00061663
Record Dates: First submitted 2018-03-23; First posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Obesity; Food Habits; Mental Depression
Keywords: obesity; food insecurity; depressive symptoms; empowerment
MeSH Terms: conditions — Obesity; Feeding Behavior; Depression; Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Intensive Intervention (Active Comparator): Three short group sessions that promote healthy lifestyles
  Interventions: Behavioral: Non-Intensive Intervention
- Intensive Intervention (Experimental): a) Individual level: a six-month intervention comprised of 12 two-hour sessions, three follow-up monthly sessions, two workshops with the participants' household members and community members and one final session that will be graduation day; b) Household level: 2 workshops about co-responsibility in the household, and self-care and nutrition, including a theater performance. Six assignments with household members' participation; c) Community level: Distribution of 2 different educational materials (one about co-responsibility and another about self-care, including healthy nutrition) and carry out the 2 workshops mentioned above, both with household and community members.
  Interventions: Behavioral: Intensive Intervention

INTERVENTIONS:
Behavioral: Intensive Intervention — an intervention focused on alleviating discouragement, food insecurity, and excess weight in women and targeted at the individual, family, and community levels
  Arms: Intensive Intervention
Behavioral: Non-Intensive Intervention — Group sessions for healthy lifestyle
  Arms: Non-Intensive Intervention

SUMMARY:
The study develops, implements, and evaluates an intervention focused on alleviating discouragement, food insecurity, and excess weight in women,targeted at the individual, family, and community levels in the Canton Central of the province of Alajuela, Costa Rica.

DETAILED DESCRIPTION:
Food insecurity is defined as "limited or uncertain availability of nutritionally adequate and safe foods or limited or uncertain ability to acquire acceptable foods in socially acceptable ways." The coexistence of excess body weight and food insecurity is recognized by researchers and increasingly by the broader public. Poverty and household food insecurity are priority topics for the global community because of their negative impacts in physical and mental health. In Costa Rica, there are no specific data about how many households are affected by food insecurity, but it is well-known that the poverty level has stood at about 20% for the past five years and that food insecurity has an economic component through material deprivation. Thus, even though food insecurity is not the same as poverty, the conditions often coexist.

Multiple studies have concluded that poverty and household food insecurity are often associated with excess body weight in women, but not men. Excess body weight, as defined as Body Mass Index ≥25, is a global health problem and the major public health problem in Costa Rican women. In 2008-2009, 59.7% of women between 20 and 44 years of age have excess body weight, reaching 77.3% in women who are 45 to 64 years of age. Excess body weight also has multiple consequences for physical and mental health. Thus, women with excess body weight and food insecurity have compromised their physical and mental health in multiple ways.

This project builds on a productive partnership between the School of Nutrition of the University of Costa Rica, the association Agenda de Mujeres, the Hospital of Alajuela, and the Women´s Office of the Municipality of Alajuela. For the last eight years, these organizations have been working together to implement health promotion interventions in low-income women with excess weight. For this project, we have the support of the University of South Carolina.

The conceptual framework that guides the intervention is based on the investigators' previous work in Costa Rica that found that discouragement - or in other words, "feeling depressed" - is the primary link in the coexistence of food insecurity and excess body weight among Costa Rican women.

The study is a 6-month intervention targeted at the individual, family, and community levels in the Canton Central of the province of Alajuela, Costa Rica. The specific aims are:

Specific Aim 1: To determine the impact of an intervention to alleviate discouragement feelings among food-insecure, excess-weight women. Hypothesis 1: After the intervention, the participants in the intervention group, as compared with the control group, will reduce their household food security status, increase their psychological and economic empowerment level, decrease their depression and anxiety levels, increase perceived social support, and decrease their body mass index and waist circumference. Qualitative methods, specifically group interviews and semi-structured in-depth interviews, also are used to assess the intervention Specific Aim 2: To qualitatively examine the impact of the intervention on gender norms, including co-responsibility in the household (i.e., joint decision-making, sharing responsibilities in the household, including taking care of children and the disabled and contributing to household support), and self-care, including healthy nutrition.

To address these aims, we designed a cluster-randomized controlled trial design at the health-center level, the first level of care in Costa Rica. Investigators randomize 15 matched pairs of health centers in a 1:1 ratio to intervention and control arms, and enroll 7 participants per health center (total n=210).

For specific aim #2 the investigators will use qualitative methods, such as group interviews, semi-structured in-depth interviews, and non-participant observation This study is significant because there are no interventions in Costa Rica or other countries that aim to improve both food security and health, including mental health and excess body weight, in food-insecure women with excess body weight. Therefore, studies are needed to develop, implement, and evaluate the efficacy and effectiveness of interventions targeting these women.

ELIGIBILITY:
Inclusion Criteria:

* Being excess weight BMI ≥ 25, according to the World Health Organization classification
* Being between 18 and 60 years old
* Being food insecure ( low, moderate, or severe) according to have a score ≥ 17 in the Food Insecurity Scale of Costa Rica
* Living in the selected community
* Being willing to participate fully in the study
* Having at least one other adult household member( ideally) or family member willing to participate

Exclusion Criteria:

* Having a diagnosis of diabetes mellitus
* Don't Know how to read and write
* Not being pregnant at the time of recruitment

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 171 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 6 months in body mass index | Baseline and 6 months
  Body mass index is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m2.
Change from baseline to 6 months in household food insecurity as assessed by the food insecurity scale for Costa Rica | Baseline and 6 months
  This scale is comprised of 14 items. The response categories include ''never,'', ''sometimes'' and ''many times."
Change from baseline to 6 months in waist circumference | Baseline and 6 months
  Waist circumference is a measure of health risk associated with excess fat around the waist.

SECONDARY OUTCOMES:
Change from baseline to 6 months in social support from family and friends for healthy eating as assessed by the social Support and Eating Habits Survey. | Baseline and 6 months
  The scale consists of 4 sub-scales
Change from baseline to 6 months in proportion of women that contribute to household support and find a job | Baseline and 6 months
  Women that began to contribute to their household support or/and found a job
Change from baseline to 6 months in psychological empowerment as assessed by the Scale of Personal Agency and Empowerment. | Baseline and 6 months
  We will use the subscale for agency of the Scale of Personal Agency and Empowerment.
Change from baseline to 6 months in the consumption of sugar drinks and fried foods as assessed by a food-frequency questionnaire | Baseline and 6 months
  We will use a food frequency with the categories: times per day, per week or per month
Change from baseline to 6 months in metabolic equivalents per week of physical activity | Baseline and 6 months
  We ask about type of activity, how many times a week and how many minutes in each session of physical activity and we will convert to metabolic equivalents per week
Change from baseline to 6 months in discouragement feelings as assessed by the Spanish version of the Hospital Anxiety and Depression Scale | Baseline and 6 months
  We will use the 7 items of the depression's subscale
Change from baseline to 6 months in anxiety symptoms as assessed by the Spanish version of the Hospital Anxiety and Depression Scale | Baseline and 6 months
  We will use the 7 items of the anxiety's subscale

CONTACTS AND LOCATIONS:
Locations (1):
- Municipality of Alajuela, Alajuela, Costa Rica

REFERENCES:
- [Background] 1. United States Department of Agriculture. Guide to Measuring Household Food Security (Revised 2000) [Internet]. [cited 2014 Oct 5]. Available from: http://www.fns.usda.gov/guide-measuring-household-food-security-revised-2000
- [Background] 2. Food Research & Action Center. Fighting Obesity and Hunger [Internet]. 2015 [cited 2015 Oct 29]. Available from: http://frac.org/initiatives/hunger-and-obesity/
- [Background] Institute of Medicine (US). Hunger and Obesity: Understanding a Food Insecurity Paradigm: Workshop Summary. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK209372/ PMID 24983070
- [Background] 4. Frongillo E, Olson C, Rauschenbach B, Kendall A. Nutritional Consequences of Food Insecurity in a Rural New York State County [Internet]. 1997 [cited 2015 Jan 6]. Available from: http://www.irp.wisc.edu/publications/dps/pdfs/dp112097.pdf
- [Background] 5. Instituto Nacional de Estadisticas y Censos. Poverty in Costa Rica [Internet]. 2014 [cited 2015 Apr 12]. Available from: http://www.inec.go.cr/Web/Home/pagPrincipal.aspx
- [Background] Schlussel MM, Silva AA, Perez-Escamilla R, Kac G. Household food insecurity and excess weight/obesity among Brazilian women and children: a life-course approach. Cad Saude Publica. 2013 Feb;29(2):219-26. doi: 10.1590/s0102-311x2013000200003. PMID 23459802
- [Background] Adams EJ, Grummer-Strawn L, Chavez G. Food insecurity is associated with increased risk of obesity in California women. J Nutr. 2003 Apr;133(4):1070-4. doi: 10.1093/jn/133.4.1070. PMID 12672921
- [Background] Townsend MS, Peerson J, Love B, Achterberg C, Murphy SP. Food insecurity is positively related to overweight in women. J Nutr. 2001 Jun;131(6):1738-45. doi: 10.1093/jn/131.6.1738. PMID 11385061
- [Background] 9. Ministerio de Salud. Encuesta Nacional de Nutrición: Fascículo Antropometría. [Internet]. 1996. Available from: http://www.binasss.sa.cr/Micro96.pdf
- [Background] Azarbad L, Gonder-Frederick L. Obesity in women. Psychiatr Clin North Am. 2010 Jun;33(2):423-40. doi: 10.1016/j.psc.2010.01.003. PMID 20385345
- [Background] 11.Martinez-Jaikel T, Frongillo E. Primary role of discouragement in co-existence of food insecurity and excess weight in Costa Rican women. J Hunger Environ Nutr. 2016;
- [Background] Gonzalez W, Jimenez A, Madrigal G, Munoz LM, Frongillo EA. Development and validation of measure of household food insecurity in urban Costa Rica confirms proposed generic questionnaire. J Nutr. 2008 Mar;138(3):587-92. doi: 10.1093/jn/138.3.587. PMID 18287371
- [Derived] Martinez-Jaikel T, Frongillo EA, Blake CE, Fram MS, Esquivel-Solis V. Reducing Both Food Insecurity and Excess Body Weight in Costa Rican Women: A Cluster Randomized Trial. Am J Prev Med. 2020 May;58(5):736-747. doi: 10.1016/j.amepre.2019.11.021. Epub 2020 Feb 6. PMID 32037021